CLINICAL TRIAL: NCT06188260
Title: Efficacy of a New Nanoemulsion Artificial Tear in Dry Eye Disease Management
Brief Title: Efficacy of a New Nanoemulsion Artificial Tear Targeting Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, LAM Chuen Thomas, FAAO, PhD, Associate Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230209004
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dry eye participants (Experimental): Participants aged 20 years or above, with OSDI score between 12-32, and with either of the following positive signs: 1) corneal staining; 2) NITBUT<10s; 3) osmolarity >=308, or difference >8
  Interventions: Drug: Systane COMPLETE Lubricant Eye Drops

INTERVENTIONS:
Drug: Systane COMPLETE Lubricant Eye Drops — Active Ingredients: Propylene Glycol 0.6% Purpose: Lubricant
  Other Names: Alcon limited

SUMMARY:
This is a prospective cohort study to compare subjective changes in symptoms using the Ocular Surface Disease Index (OSDI) questionnaire, following the recommended dosage of the new nanoemulsion eye drops (Systane Complete)in mild to moderate dry eye patients, and to investigate objective ocular surface changes using modern clinical instruments during the study period.

DETAILED DESCRIPTION:
This study, lasting for 3 months in total, is to investigate the changes in both subjective reports (OSDI score) and objective measurements (Non-invasive Tear Break Time (NITBUT) and other clinical signs such as corneal staining) after the use of this nanoemulsion eye drops (Systane Complete). Subjects are required to use the eyedrop qid for 3 months, and come back for follow-up at 2-week and 3-month visits. Other secondary measurements such as Meibography and lipid layer thickness, will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-50 years old
2. Best corrected distance visual acuity ≥ 6/9
3. Mild to moderate OSDI score 13-32
4. Any one of the objective test positive (NITBUT/Corneal fluorescein staining/Tear osmolarity)

Exclusion Criteria:

1. Any active ocular infections
2. Inflammations or anomalies in the eyelid
3. Uncontrolled, newly diagnosed systemic diseases or with modified long-term medications within 6 months that are known to affect tear profile.
4. Pregnancy and breastfeeding
5. Contact lens wearers are required to stop contact lenses wear for at least 1 week before the evaluation.
6. Subjects who are using artificial tears or other eyedrops will be excluded.
7. Subjects who are taking systemic drugs that may cause dry eye, e.g., Antidepressants/antipsychotics, Systemic corticosteroids.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Change in OSDI score at 2-week visit
  Change in OSDI score at 2-week visit

SECONDARY OUTCOMES:
Non invasive tear break-up time (NITBUT) | NITBUT at 2-week and 3-month visits
  NITBUT at 2-week and 3-month visits
Meibography | Meibography at 2-week and 3-month visits
  Meibography at 2-week and 3-month visits

CONTACTS AND LOCATIONS:
Overall Officials: Thomas LAM, PhD, Principal Investigator — The Hong Kong Polytechnique University
Locations (1):
- Thomas LAM, Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Liao X, Guo B, Bian J, Li PH, Tse JSH, Ngo W, Zhou L, Lam T. Efficacy of a new nanoemulsion artificial tear in dry eye disease management: Study protocol for a prospective cohort study. PLoS One. 2025 May 9;20(5):e0323523. doi: 10.1371/journal.pone.0323523. eCollection 2025. PMID 40343954